CLINICAL TRIAL: NCT03810274
Title: 3DV+TPS Software Outlines the Outline of Radiotherapy for Nasopharyngeal Carcinoma Center Comparison Study Clinical Research
Brief Title: 3DV+TPS Software Outlines the Radiotherapy of Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy Director, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-012
Record Dates: First submitted 2019-01-11; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Radiotherapy; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3DV+TPS: This experiment included a total of 300 patients with nasopharyngeal carcinoma, using 3DV + TPS software and imported TPS, domestic TPS, these three sets of TPS delineate bilateral crystal, bilateral optic nerve, bilateral eyeball, bilateral parotid gland, oral cavity, spinal cord There are 12 organs in the brainstem and brain, and the accuracy and speed of the 3 sets of TPS sketches are compared.
  Interventions: Device: 3DV+TPS；VARIAN TPS；FonicsPlan

INTERVENTIONS:
Device: 3DV+TPS；VARIAN TPS；FonicsPlan

SUMMARY:
Comparing the accuracy and speed of 3DV+TPS software with imported TPS and domestic TPS to outline the contours of crisis organs, it is proved that 3DV+TPS has superiority compared with domestic TPS, and it has non-inferiority compared with imported TPS, indicating that the software can improve contour sketching accuracy. And speed, reduce the burden on doctors, improve medical efficiency.

DETAILED DESCRIPTION:
Comparing the accuracy and speed difference between 3DV+TPS software and imported TPS and domestic TPS to outline the contours of crisis organs, the selected organs are: bilateral eyeballs, bilateral crystals, bilateral optic nerves, bilateral parotid glands, oral cavity, spinal cord, brainstem, The brain has a total of 12 organs; verify that 3DV+TPS is superior to domestic TPS, and has non-inferiority compared with imported TPS, Ming software can improve the accuracy and speed of contour sketching, reduce the burden on doctors, and improve medical efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. It is diagnosed as nasopharyngeal carcinoma by histopathological examination, and there is no tumor invasion in the organs that need to be assessed;
2. Age 18-70 years old;
3. There is nasopharynx localization enhanced CT, nasopharynx enhanced MRI.

Exclusion Criteria:

1. Patient information is incomplete; no age, gender, MRI, height, radiotherapy location CT;
2. The organs at risk that need to be assessed are invaded by the tumor;
3. Any reason cannot be combined with the research or the researcher believes that it is not suitable for inclusion in this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 7 different grade hospital radiotherapy centers have received radiotherapy for patients with nasopharyngeal carcinoma Case information, based on inclusion and exclusion criteria, a total of 300 cases were screened. Among them, Xinqiao Hospital collected 180 cases, He collected 20 cases in 20 hospitals, totaling 200 cases.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Sketching accuracy | one year
  Define ΔV as a percentage of the total volume of the gold standard;
Sketch speed | one year
  Use the stopwatch to record the total time used to draw down 12 organs, to start sketching as the starting point of the time, and to finish the saving of the data.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China